CLINICAL TRIAL: NCT06914635
Title: Immunotherapy: Care and Prevention of Infectious and Tumoral Diseases (ImmunoHUB)
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Mario Mondelli, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: 0047354/23
Record Dates: First submitted 2025-03-21; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: SARS CoV-2; Liver Tumours
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Recovered subjects after SARS-CoV-2 infection
- Patients with primary liver tumor.

SUMMARY:
The project comprises two research lines. In the line 1, human monoclonal antibodies toward SARS-CoV-2 will be generate and characterized by in vitro functional tests. In the line 2, in vitro tests will be performed to evaluate the efficency of immune response mediated by antibodies direct to specific tumor molecules.

ELIGIBILITY:
Inclusion Criteria:

Line 1: - Age >18 at time of signing informed consent form

* Signed informed consent form Line 2: - Primery liver tumor
* Age >18 at time of signing informed consent form
* Signed informed consent form

Exclusion Criteria:

Line 1: - Active or history of neoplastic malignancy

* Active autoimmune disease ongoing treatment with immunosuppressive therapy
* Evidence of positive HIV, HCV, HBV test
* Diabetes
* Failure to sign informed consent form Line 2: - Concomitant diseases with life expectancy of less than 12 months
* Chronic autoimmune or inflammatory diseases
* Treatment with atezolizumab, bevacizumab, sorafenib, lenvatinib, regorafenib, cabozantinib, checkpoint inhibitors and tyrosine kinase inhibitors or anti-VEGF therapies
* Other extrahepatic neoplasms occurring or in the last 3 years except for tumors resected with curative intent and without evidence of relapse for >3 years prior to signing informed consent and considered low risk of relapse
* HIV infection
* Failure to sign informed consent form

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Line 1: Recovered subjects from SAS-CoV-2 infection. Line 2: Patients with primary liver tumor
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2025-02-19 (Actual); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
The efficiency of antibodies will be evaluated toward SARS-CoV-2 and liver primary tumor cells by functional in vitro tests. | From enrollement to 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia, Pavia, Italy